CLINICAL TRIAL: NCT05414305
Title: The Female Microbiome in Patients Undergoing Bladder Instillation Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Collaborators: US Army Medical Research Institute of Infectious Diseases (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: WRNMMC-EDO-2021-0728
Record Dates: First submitted 2022-05-26; First posted 2022-06-10 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Interstitial Cystitis; Bladder Pain Syndrome; Microbial Colonization
MeSH Terms: conditions — Cystitis, Interstitial; Communicable Diseases | interventions — Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Heparin & Alkalinized Lidocaine Bladder Instillation (Other): Six weekly bladder instillations, each instillation consisting of 40,000 IU Heparin, 200mg lidocaine, 2ml 8.4% sodium bicarbonate, sterile water for a total volume 50 milliliters (mL).
  Interventions: Drug: Heparin & Alkalinized Lidocaine Bladder Instillation

INTERVENTIONS:
Drug: Heparin & Alkalinized Lidocaine Bladder Instillation — Bladder instillation instilled via catheter and to dwell for minimum of 30 minutes prior to spontaneous void

SUMMARY:
The underlying pathophysiology for BPS/IC is currently an active area of research. There is speculation that there may be alteration in the bladder and vaginal microbiome that contributes to the symptomatology of BPS/IC, however existing literature is limited and contradictory. Nickel et al (2015) studied the bladder microbiota in women with IC/BPS during a flare versus nonflare. The study collected initial stream and midstream urine specimens and detected overall, there was no significant differences in the species composition. However, a greater prevalence of fungi (Candida and Saccharomyces) was seen in the flare group (15.7%) versus the non-flare group (3.9%) midstream urine specimens. Pearce et al (2015) sought to characterize the urinary microbiome via catheterized specimens from women with urgency urinary incontinence, a condition that can present similarly as IC/BPS. The study found that more than half of the patients were sequence positive, most commonly for Lactobacillus (45%) or Gardnerella (17%), with 25% made up of various other bacteria. In contrast, Abernethy et al (2017) showed via catheterized urine specimens from patients with IC/BPS that the urinary microbiome is less diverse and less likely to contain Lactobacillus species. There have been two recent studies investigating the female urinary microbiome in patients with IC/BPS. Nickel et al (2019) found no differences in species composition between urine from patients with IC/BPS versus controls. Meriwether et al (2019) reported similar findings, and additionally found no differences when comparing the vaginal bacterial microbiome in patients with IC/BPS versus controls. However, in evaluating the bladder microbiome, both studies utilized uncatheterized urine specimens. Wolfe et al (2012) showed microbiome differences between clean-catch and catheterized urine specimens, therefore vaginal contamination in both studies cannot be ruled out.

DETAILED DESCRIPTION:
This study uses samples collected under an interventional study and consented for use in future research - this study is use of those samples under the future research provision, and this study was deemed to meet exempt category 4.

ELIGIBILITY:
Inclusion Criteria:

* Patients who previously or will be undergoing bladder instillation therapy for treatment of IC/BPS and whom had or will have urine/vaginal specimens collected at the beginning and between 4-6th instillations.

Exclusion Criteria:

* Patients not meeting inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Change of the female microbiome as measured by bacterial ribosomal RNA sequencing in patients with BPS/IC at baseline and during bladder instillation therapy | Baseline, 4-6 weeks

SECONDARY OUTCOMES:
Correlation of female microbiome as measured by bacterial ribosomal RNA sequencing and O'Leary-Sant questionnaire scores | Baseline, 4-6 weeks
  Consists of O'Leary-Sant Symptom and Problem Index. Total score 0-36, with higher scores indicating worse symptoms
Correlation of female microbiome as measured by bacterial ribosomal RNA sequencing and Female Sexual Function Index (pain) questionnaire scores | Baseline, 4-6 weeks
  Total score 0-6, with higher scores indicating worse symptoms
Correlation of female microbiome as measured by bacterial ribosomal RNA sequencing and Female Sexual Distress-Revised Inventory questionnaire scores | Baseline, 4-6 weeks
  FSDS-R evaluates distress associated with inadequate/impaired sexual function. Total score 0-52, with higher scores indicating worse symptoms
Correlation of female microbiome as measured by bacterial ribosomal RNA sequencing and Short Form 12 questionnaire scores | Baseline, 4-6 weeks
  SF-12 is a general health questionnaire that evaluates quality of life measures, divided into mental and physical component scores. Higher scores associated with better symptoms.
Correlation of female microbiome as measured by bacterial ribosomal RNA sequencing and Visual Analog Scale questionnaire scores | Baseline, 4-6 weeks
  Scale of 0-10 (0= no pain, 10 = worst pain)
Characterization of bacterial species present as measured by bacterial ribosomal RNA sequencing in the vaginal and urinary microbiome | Baseline, 4-6 weeks
Characterization of bacterial species diversity as measured by bacterial ribosomal RNA sequencing in the vaginal and urinary microbiome | Baseline, 4-6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eva K Welch, MD MS, Principal Investigator — Walter Reed National Military Medical Center
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wolfe AJ, Toh E, Shibata N, Rong R, Kenton K, Fitzgerald M, Mueller ER, Schreckenberger P, Dong Q, Nelson DE, Brubaker L. Evidence of uncultivated bacteria in the adult female bladder. J Clin Microbiol. 2012 Apr;50(4):1376-83. doi: 10.1128/JCM.05852-11. Epub 2012 Jan 25. PMID 22278835
- [Background] Pearce MM, Zilliox MJ, Rosenfeld AB, Thomas-White KJ, Richter HE, Nager CW, Visco AG, Nygaard IE, Barber MD, Schaffer J, Moalli P, Sung VW, Smith AL, Rogers R, Nolen TL, Wallace D, Meikle SF, Gai X, Wolfe AJ, Brubaker L; Pelvic Floor Disorders Network. The female urinary microbiome in urgency urinary incontinence. Am J Obstet Gynecol. 2015 Sep;213(3):347.e1-11. doi: 10.1016/j.ajog.2015.07.009. Epub 2015 Jul 23. PMID 26210757
- [Background] Abernethy MG, Rosenfeld A, White JR, Mueller MG, Lewicky-Gaupp C, Kenton K. Urinary Microbiome and Cytokine Levels in Women With Interstitial Cystitis. Obstet Gynecol. 2017 Mar;129(3):500-506. doi: 10.1097/AOG.0000000000001892. PMID 28178051
- [Background] Meriwether KV, Lei Z, Singh R, Gaskins J, Hobson DTG, Jala V. The Vaginal and Urinary Microbiomes in Premenopausal Women With Interstitial Cystitis/Bladder Pain Syndrome as Compared to Unaffected Controls: A Pilot Cross-Sectional Study. Front Cell Infect Microbiol. 2019 Apr 8;9:92. doi: 10.3389/fcimb.2019.00092. eCollection 2019. PMID 31024861
- [Background] Nickel JC, Stephens-Shields AJ, Landis JR, Mullins C, van Bokhoven A, Lucia MS, Henderson JP, Sen B, Krol JE, Ehrlich GD; MAPP Research Network. A Culture-Independent Analysis of the Microbiota of Female Interstitial Cystitis/Bladder Pain Syndrome Participants in the MAPP Research Network. J Clin Med. 2019 Mar 26;8(3):415. doi: 10.3390/jcm8030415. PMID 30917614
- [Background] Nickel JC, Stephens A, Landis JR, Mullins C, van Bokhoven A, Lucia MS, Ehrlich GD; MAPP Research Network. Assessment of the Lower Urinary Tract Microbiota during Symptom Flare in Women with Urologic Chronic Pelvic Pain Syndrome: A MAPP Network Study. J Urol. 2016 Feb;195(2):356-62. doi: 10.1016/j.juro.2015.09.075. Epub 2015 Sep 26. PMID 26410734